CLINICAL TRIAL: NCT01654042
Title: Prolongation of the Interval Between Prothrombin Time Tests in Stable Patients II (the PRINT II Study): a Randomized Controlled, Non-inferiority Trial Comparing 4-weekly With 12-weekly Testing and Dose-assessment
Brief Title: Prolongation of the Interval Between Prothrombin Time Tests in Stable Patients II
Acronym: PRINT-II
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No funding obtained
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sam Schulman, SSchulman, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRINT-II-2012
Record Dates: First submitted 2012-07-21; First posted 2012-07-31 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Atrial Fibrillation; Valvular Heart Disease; Deep Vein Thrombosis; Pulmonary Embolism; Peripheral Arterial Disease
Keywords: anticoagulation; warfarin; monitoring; bleeding; thromboembolism
MeSH Terms: conditions — Atrial Fibrillation; Heart Valve Diseases; Venous Thrombosis; Pulmonary Embolism; Peripheral Arterial Disease; Hemorrhage; Thromboembolism | interventions — International Normalized Ratio

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard interval between PT testing (No Intervention): Prothrombin time (PT) is tested every 4 weeks, according to American College of Chest Physicians (ACCP) Guidelines up to 2008 for stable patients on warfarin.
- Prolonged interval between PT testing (Experimental): Prothrombin time (PT) is tested every 12 weeks, according to suggestion in American College of Chest Physicians (ACCP) Guidelines of 2012 for stable patients on warfarin.
  Interventions: Other: Prolonged interval between PT testing

INTERVENTIONS:
Other: Prolonged interval between PT testing — Patients in the intervention group will be scheduled for prothrombin time testing and dosing of warfarin every 12 weeks instead of every 4 weeks. This has been suggested in the latest edition of the ACCP guidelines as a possibility for very stable patients. In order to change this from a suggestion to a formal recommendation a study powered for clinically important outcomes is needed.
  Other Names: INR (International Normalized Ratio) tests
  Arms: Prolonged interval between PT testing

SUMMARY:
More than 2 million patients in North America are treated with warfarin - a "blood thinner" - to prevent blood clots in arteries or veins. The treatment has to be monitored with a blood test and the dose changed accordingly every 1-4 weeks. One third of the patients have very stable results and hardly ever have to change the dose. The investigators wish to show that the level of control of the treatment with warfarin in these very stable patients is not worse with 12-weekly testing. A pilot study the investigators performed indicated that 12-weekly testing would be safe but this has to be confirmed in a large study. One third of patients taking warfarin have not had any changes in the dose for the past 6 months or longer. These patients will be asked about participation in the study. They will be randomized to testing and dosing every 4 or 12 weeks. Each patient is in the study until it ends, which will be minimum 1 year and can be up to about 4 years. The study is designed to show that 12-weekly testing does not significantly increase the risk for major bleeding or blood clots. The results would be important for a large number of patients. An increase of the interval between blood tests from 4 to 12 weeks would reduce the burden for these patients on life-long treatment considerably.

DETAILED DESCRIPTION:
The study is a randomized, controlled, open-label, multi-center non-inferiority trial to demonstrate that the interval between internation normalized ration (INR) tests can be extended from the recommended 4 weeks to 12 weeks for patients with stable INRs. PROBE design. Patients receiving warfarin therapy that have exhibited INR stability, defined as no change in maintenance dose for at least 6 months, are potentially eligible for enrolment in the study. The primary outcome is a composite of major bleeding (ISTH criteria) plus objectively verified arterial or venous thromboembolism (excluding superficial thrombophlebitis) plus death related to thromboembolism. Justification: the study is not reflecting a "trade-off" scenario where one regimen is expected to be more effective at the cost of increased harm compared to the other regimen. Conversely, the potential disadvantage of the experimental regimen in this trial is increased variability in INR, which may result in an increased rate of low as well as high INRs and therefore potentially an increase of both types of clinical events.

ELIGIBILITY:
Inclusion Criteria:

* long-term warfarin for prophylaxis of arterial embolism due to atrial fibrillation or mechanical heart valve replacement OR secondary prophylaxis after VTE
* therapeutic INR range of 2.0-3.0 or 2.5-3.5
* anticoagulation therapy has been managed by the study site for at least 6 months prior to enrollment
* warfarin maintenance dose has remained unchanged for the previous 6 months or longer

Exclusion Criteria:

* Age < 18 years
* Life expectancy of less than 1 year
* Congestive heart failure or other diagnosis where the condition or its treatment is expected to affect the stability of INR (e.g. cancer requiring chemotherapy)
* Attending physician believes that patient is not suitable for the study (for instance, psychiatric disorder; history of non-compliance; newly diagnosed disease which by itself, via the treatment required or the effects thereof may cause instability of INRs)
* Patients who perform self-testing
* Geographic inaccessibility
* Failure to obtain written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Composite of major bleeding and objectively verified arterial or venous thromboembolism | Average 3 years
  The justification for a composite outcome including both bleeding and thromboembolism is that the study is not reflecting a "trade-off" scenario where one regimen is expected to be more effective at the cost of increased harm compared to the other regimen. Conversely, the potential disadvantage of the experimental regimen in this trial is increased variability in prothrombin time, which may result in an increased rate of short as well as long prothrombin times and therefore potentially an increase of both types of clinical events.

SECONDARY OUTCOMES:
All-cause mortality | Average 3 years
Any bleeding | Average 3 years
  This is the composite of major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schulman, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Schulman S, Parpia S, Stewart C, Rudd-Scott L, Julian JA, Levine M. Warfarin dose assessment every 4 weeks versus every 12 weeks in patients with stable international normalized ratios: a randomized trial. Ann Intern Med. 2011 Nov 15;155(10):653-9, W201-3. doi: 10.7326/0003-4819-155-10-201111150-00003. PMID 22084331
- [Background] Pengo V, Barbero F, Biasiolo A, Pegoraro C, Cucchini U, Iliceto S. A comparison between six- and four-week intervals in surveillance of oral anticoagulant treatment. Am J Clin Pathol. 2003 Dec;120(6):944-7. doi: 10.1309/U716-4E0X-H5UE-RKRV. PMID 14671984